CLINICAL TRIAL: NCT05186233
Title: Innovations in Wearable Technology for Correcting Circadian Misalignment in Shift Work Disorder
Brief Title: Use of Consumer Sleep Technology to Treat Shift Work Disorder
Acronym: SHIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Philip Cheng, Assistant Scientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15108
Record Dates: First submitted 2021-12-15; First posted 2022-01-11 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2024-09

CONDITIONS: Shift-work Disorder
MeSH Terms: interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-personalized light condition (Active Comparator): Participants will receive light exposure recommendations from the SHIFT mobile application based on their habitual sleep schedule. Participants will follow these recommendations over the course of two weeks.
  Interventions: Behavioral: Phototherapy
- Personalized light condition (Experimental): Participants will receive light exposure recommendations from the SHIFT mobile application based on their activity levels. Participants will follow these recommendations over the course of two weeks.
  Interventions: Behavioral: Phototherapy

INTERVENTIONS:
Behavioral: Phototherapy — Light exposure recommendations provided by SHIFT mobile application

SUMMARY:
The purpose of this study is to examine the effectiveness of a personalized light exposure schedule for Shift Work Disorder (SWD) in night shift workers compared to a non-personalized light exposure schedule.

DETAILED DESCRIPTION:
Participants will be randomized into each condition (n = 25) in a 1:1 ratio. Variables of interest, dim light melatonin onset (DLMO) and shift work disorder (SWD) symptoms, will be assessed before and after the intervention, which will last two weeks. All participants (N=50) will be asked to wear an Apple Watch for two weeks leading up to an in-lab visit. Activity data collection from the Apple Watch will be processed through a mathematical model of the human circadian pacemaker (previously validated in SWD) to generate estimates of DLMO. This two-week period is followed by a 27-hour laboratory visit for pre-treatment assessment of DLMO (hourly saliva melatonin samples over 24 hours). At the end of this visit, participants will receive an orientation to the SHIFT mobile application, where they will be able to assess their prescribed light exposure schedule.

ELIGIBILITY:
Inclusion Criteria:

* Participants must work at least 2 night shifts a week
* Participants must have night shifts starting between 18:00 and 02:00 and lasting 8 to 12 hours
* Participants must have maintained this night shift schedule for at least 6 months
* Participants must have Shift Work Disorder, diagnosed based on ICSD-3 criteria

Exclusion Criteria:

* Medical history of central nervous system disorders
* Medical history of other sleep disorders
* Diagnosis of an unstable major medical condition medical chart review
* Dependence on alcohol (≥ 4 beverages a day)
* Heavy tobacco use (≥ 10 cigarettes per day)
* Recreational drug use
* Use of medications impacting central nervous system functioning
* Caffeine use in excess of 5-6 servings (~ 600mg) per day
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Dim light melatonin onset | Within two days of treatment for a duration of 24 hours
  Melatonin values will be measured in saliva samples, collected in dim light conditions in a laboratory, to determine circadian phase.

SECONDARY OUTCOMES:
Insomnia | Within one week of post-treatment
  Insomnia will be measured with the Insomnia Severity Scale (0 to 28; higher scores correspond to worse severity)
Daytime sleepiness | Within one week of post-treatment
  Sleepiness will be measured with the Epworth Sleepiness Scale (0 to 24; a score of 10 or greater indicates excessive daytime sleepiness)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Columbus Medical Center, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Request for data sharing will be evaluated on a case-by-case basis.